CLINICAL TRIAL: NCT04179864
Title: CELLO-1: A Phase 1b/2 Open-Label Study Evaluating Tazemetostat in Combination With Enzalutamide or Abiraterone/Prednisone in Chemotherapy Naive Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of Tazemetostat With Enzalutamide or Abiraterone/Prednisone in Participants With Advanced Prostate Cancer
Acronym: CELLO-1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision, no safety concern
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EZH-1101; 2019-003649-14 (EudraCT Number)
Record Dates: First submitted 2019-11-14; First posted 2019-11-27 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
Keywords: metastatic castration resistant prostate cancer; tazemetostat; EPZ-6438; E7438; enzalutamide; abiraterone; Prednisone; Zytiga; Xtandi
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tazemetostat; abiraterone; Prednisone; Abiraterone Acetate; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1b: Tazemetostat in Combination with Abiraterone/Prednisone (Experimental): In Phase 1b, abiraterone/prednisone will be administered in combination with tazemetostat in cycle 1 (28 days) to establish the recommended dose of tazemetostat in this combination; participants may continue treatment in additional 28-day cycles, as tolerated, until progression or unacceptable toxicity
  Interventions: Drug: Tazemetostat; Drug: Abiraterone/prednisone
- Phase 1b: Tazemetostat in Combination with Enzalutamide (Experimental): In Phase 1b, enzalutamide will be administered in combination with tazemetostat in cycle 1 (28 days) to establish the recommended dose of tazemetostat in this combination; participants may continue treatment in additional 28-day cycles, as tolerated, until progression or unacceptable toxicity
  Interventions: Drug: Tazemetostat; Drug: Enzalutamide
- Phase 2: Tazemetostat in Combination with Enzalutamide (Experimental): Participants will receive the newly established recommended phase 2 dose, orally twice daily when given in combination with enzalutamide) as determined in phase 1b part of the study) or enzalutamide alone.
  All participants will receive treatment in 28-day cycles.
  Interventions: Drug: Tazemetostat; Drug: Enzalutamide
- Phase 2: Enzalutamide only (Active Comparator): In Phase 2, Enzalutamide will be administered on cycle 1 day 1
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Tazemetostat — Tazemetostat (EPZ-6438) is a selective small-molecule inhibitor of the histone-lysine methyltransferase EZH2 gene
  Other Names: EPZ-6438; E7438; IPN60200
  Arms: Phase 1b: Tazemetostat in Combination with Abiraterone/Prednisone; Phase 1b: Tazemetostat in Combination with Enzalutamide; Phase 2: Tazemetostat in Combination with Enzalutamide
Drug: Abiraterone/prednisone — 1,000 mg (two 500 mg tablets or four 250 mg tablets) orally once daily in combination with prednisone 5 mg administered orally twice daily.
  Other Names: Zytiga
  Arms: Phase 1b: Tazemetostat in Combination with Abiraterone/Prednisone
Drug: Enzalutamide — enzalutamide 160 mg (four 40 mg capsules) orally once daily
  Other Names: Xtandi
  Arms: Phase 1b: Tazemetostat in Combination with Enzalutamide; Phase 2: Enzalutamide only; Phase 2: Tazemetostat in Combination with Enzalutamide

SUMMARY:
This is a global, multi-center, open-label, randomized phase 1b/2, active-controlled safety and efficacy study of oral administration of tazemetostat in combination with enzalutamide or abiraterone/prednisone (phase 1b) versus enzalutamide or abiraterone/prednisone alone in asymptomatic or mildly symptomatic subjects with progressive, metastatic castration-resistant prostate cancer (mCRPC) who have progressed on either abiraterone acetate, enzalutamide, or apalutamide or who are second generation anti-androgen treatment naive, and who have not received chemotherapy for mCRPC.

This study is designed to determine the recommended phase 2 doses (RP2D) of tazemetostat in combination with either enzalutamide or abiraterone/prednisone, based on safety, tolerability, pharmacokinetic, pharmacodynamic, and efficacy profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of consent ≥ 18 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 (Appendix
3. Life expectancy of > 3 months.
4. Histologically or cytologically confirmed adenocarcinoma of the prostate. Small cell or neuroendocrine tumors of the prostate are also permitted.
5. Progressive disease in the setting of medical or surgical castration (ie, castration- resistant prostate cancer [CRPC]) by PCWG3 criteria for study entry.

   * Evidence of disease progression by rising PSA or
   * Soft tissue progression per RECIST 1.1 or
   * Evidence of disease progression by observation of 2 new bone lesions since the initiation of last systemic therapy.
6. Metastatic prostate cancer disease, documented by the following imaging

   • Bone lesions on bone scan (per PCWG3) or by soft tissue disease (per RECIST 1.1) by CT/MRI imaging Must have undergone bilateral orchiectomy or be willing to continue GnRH analogue or antagonist.
7. Prior treatment with a second-generation androgen inhibitor as follows:

   * For phase 1b, EITHER Previously untreated with or progressed on a second generation androgen inhibitor (abiraterone, enzalutamide, or apalutamide) OR progressed on a second generation inhibitor (inhibitor (abiraterone, enzalutamide, or apalutamide)
   * For phase 2 randomized component (i.e, enzalutamide- containing treatment arms) of the study, previously progressed on abiraterone.

Exclusion Criteria:

1. Known symptomatic brain metastases
2. Treatment with any of the following for prostate cancer within the indicated timeframe prior to day 1 of starting study treatment:

   * First generation: AR antagonists (eg, bicalutamide, nilutamide, flutamide) within 4 weeks.
   * 5-alpha-reductase inhibitors, ketoconazole, estrogens (including diethylstilbesterol), or progesterones within 2 weeks.
   * Chemotherapy (except as permitted in inclusion criteria #10) within 3 weeks.
   * Prior radionuclide therapy within 4 weeks.
   * Another interventional product or standard agent in a clinical study within 28 days prior to the first planned dose of Tazemetostat
   * For phase 2 subjects to be randomized to one of the enzalutamide treatment arms only, prior treatment with the second-generation androgen antagonist including enzalutamide, apalutamide, darolutamide, and proxalutamide, etc.
3. Severe concurrent disease, infection, or comorbidity that, in the judgment of the Investigator, would make the subject inappropriate for enrollment
4. Has had prior exposure to tazemetostat or other inhibitor(s) of enhancer of zeste homologue-2.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Ph 1b: Percentage of Participants with Treatment Emergent Adverse Event (TEAEs) | At end of Cycle 1 (each cycle is 28 days)
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Ph 1b: Select the recommended phase 2 doses (RP2D) of tazemetostat for each combination | 1 cycle/28 days
  Based on pharmacokinetic (PK) and pharmacodynamic parameters as well as efficacy and the overall tolerability of each of the combinations (tazemetost with enzalutamide or tazemetostat with abiraterone/prednisone)
Ph 2: Change in radiographic progression free survival (rPFS) | Day 1 of Cycles 3, 5, 7, 10, and 13, and every 12 weeks after Cycle 13 for 1 year (each cycle is 28 days)
  Assessed by change radiographic progression free survival (rPFS) according to Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria for progression in bone or in soft tissue

SECONDARY OUTCOMES:
Phase 1b and 2: Percentage of participants with a ≥50% decline of Prostate Specific-Antigen (PSA50). | From baseline at any time on study, an average of one year
  For participants with a baseline PSA ≥2.0 ug/L (ng/mL) per PCWG3 criteria
Phase 1b and 2: Objective response rate (ORR) and best overall response (BOR) in soft tissue | At 6 months on treatment.
  According to Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) guidelines.
Phase 1b and 2: Disease control rate (DCR) | At 6 months on treatment.
  Assessed by radiographic progression per PCWG3 criteria, with no unequivocal clinical progression or death
Phase 1b and 2: Time to first skeletal-related event (SRE) | During screening and every 9 weeks if clinically indicated at baseline, average of one year
Phase 1b and 2: Time to initiation of the next systemic treatment for prostate cancer (TTNT) | From baseline to end of study, an average of one year
  TTNT is defined as the time from the date of randomization to date of first documented administration of the next systemic treatment for prostate cancer.
Phase 1b and 2: Time to PSA progression (TTPP) | From baseline to the day of PSA progression, an average one one year.
  Defined as the duration per PCWG3 criteria in months.
Phase 1b and 2: Reduction in circulating tumor cells (CTC) | From screening to 30 days after last dose
  From a state of having a detectable number of CTCs to having an undetectable number of CTCs
Phase 1b and 2: CTC response rate | From baseline to end of study, an average of one year
  Defined as the percentage of participants with a ≥30% reduction in CTC number
Phase 1b and Phase 2: Percentage of Participants with Treatment Emergent Adverse Event (TEAEs) | From baseline to end of study, an average of one year
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Phase 1b and 2: AUC0-last: area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration. | From baseline to end of study, an average of one year
  AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Phase 1b and 2:AUC0-24: area under the plasma concentration-time curve from time 0 to the time of 24 hours. | From baseline to end of study, an average of one year
  AUC_0-24 is defined as the concentration of drug over time from time zero to 24 hours.
Phase 1b and 2: Cmax: maximum plasma concentration. | From baseline to end of study, an average of one year
  Cmax is defined as the maximum observed concentration of drug.
Phase 2: Change in Functional Assessment of Cancer Therapy - Prostate (FACT-P) | From baseline to end of study, an average of one year
  Assessed by Well-being Subscale (FWB) and Prostate Cancer Subscale (PCS) scores
Phase 2: Time to definitive deterioration (TDD) in functional status and in prostate symptoms | From baseline to end of study, an average of one year
  Assessed by the FACT-P FWB and PCS scores.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (24):
- United States (16):
  - Genesis Healthcare Partners, San Diego, California
  - The Urology Center Of Colorado, Denver, Colorado
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - XCancer - Northwest Oncology and Hematology, Rolling Meadows, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Associated Medical Professionals of NY, PLLC - Urology, Syracuse, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - University of Pittsburgh Medical Center - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - SCRI - Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Urology Associates P.C., Hendersonville, Tennessee
  - XCancer - Tennesee Cancer Specialists, Knoxville, Tennessee
  - SCRI - Tennessee Oncology Nashville, Nashville, Tennessee
  - Urology San Antonio, San Antonio, Texas
- Academisch Ziekenhuis Groeninge Campus Kennedylaan, Kortrijk, West Vlaanderen, Belgium
- Spain (7):
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera, Cadiz
  - Hospital de la Santa Creu i. Sant Pau, Barcelona
  - Hospital del Mar Parc de Salut Mar, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: http://vivli.org/members/ourmembers/